CLINICAL TRIAL: NCT00003808
Title: Phase II Study of Theophylline in Chronic Lymphocytic Leukemia
Brief Title: Theophylline in Treating Patients With In Situ, Stage I, or Stage II Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network)
Purpose: Treatment
Other Study IDs: CDR0000066953; E-4998; NCCTG-988151
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Theophylline

INTERVENTIONS:
Drug: theophylline

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of theophylline in treating patients who have in situ, stage I, or stage II chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in asymptomatic patients with stage 0, I, or II B-cell chronic lymphocytic leukemia treated with theophylline. II. Determine the toxicity of this treatment in these patients.

OUTLINE: Patients receive oral theophylline daily. Daily treatment continues for a maximum of 6 months in the absence of disease progression or unacceptable toxicity. Patients are followed every 4 months for 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study over approximately 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage 0, I, or II B-cell chronic lymphocytic leukemia Stable disease that would otherwise be observed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 1 year Hematopoietic: Absolute lymphocyte count greater than 5,000/mm3 Mature lymphocytes with less than 55% prolymphocytes, atypical lymphocytes, or lymphoblasts Bone marrow with at least 30% lymphocytes Hepatic: No cirrhosis Renal: Not specified Cardiovascular: No history of unstable cardiac arrhythmia No active congestive heart failure Other: No history of uncontrolled seizure disorder Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent condition that would make life expectancy less than 1 year

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent interferon alfa Chemotherapy: No prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 3 months since prior corticosteroids No concurrent corticosteroids Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08-11 (Actual); Primary Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Della Makower, MD, Study Chair — Albert Einstein College of Medicine; Rajiv K. Pruthi, MBBS, Study Chair — Mayo Clinic
Locations (71):
- United States (68):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - Kaplan Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Wiernik PH, Paietta E, Goloubeva O, Lee SJ, Makower D, Bennett JM, Wade JL, Ghosh C, Kaminer LS, Pizzolo J, Tallman MS; Eastern Cooperative Oncology Group. Phase II study of theophylline in chronic lymphocytic leukemia: a study of the Eastern Cooperative Oncology Group (E4998). Leukemia. 2004 Oct;18(10):1605-10. doi: 10.1038/sj.leu.2403494. PMID 15356646